CLINICAL TRIAL: NCT06661252
Title: Evaluation of Nasal Biomarkers for Objective Assessment of Disease Severity in Respiratory Disorders
Acronym: ENBOARD
Status: Recruiting | Type: Observational
Sponsor: Diag-Nose Medical Pty Ltd (Other)
Responsible Party: Sponsor
Other Study IDs: DNM_002_V240930
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma Patients; Asthma and Rhinitis; Asthmatic Patients; Asthma, Chronic Obstructive Pulmonary Disease (COPD); Rhinitis Allergic; Rhinitis, Allergic, Perennial and/or Seasonal; Non-allergic Rhinitis; Chronic Sinusitis With or Without Nasal Polyps; Healthy Volunteers
Keywords: Nasal biomarker; Nasal fluid; Asthma biomarker; COPD biomarker; Rhinitis biomarker; Chronic sinusitis biomarker; Allergy; Respiratory disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Rhinitis; Rhinitis, Allergic, Perennial; Common Cold; Hypersensitivity; Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal fluid samples will be collected using the ABEL microsampler device.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (5):
- Healthy Controls: Healthy volunteers.
  Interventions: Device: ABEL microsampler device
- COPD sufferers: Previously diagnosed COPD sufferers.
  Interventions: Device: ABEL microsampler device
- Asthma sufferers: Previously diagnosed asthma sufferers of various subtypes.
  Interventions: Device: ABEL microsampler device
- Allergic rhinitis sufferers: Previously diagnosed seasonal or perennial allergic rhinitis sufferers.
  Interventions: Device: ABEL microsampler device
- Chronic sinusitis sufferers: Previously diagnosed chronic sinusitis sufferers with/without nasal polyps.
  Interventions: Device: ABEL microsampler device

INTERVENTIONS:
Device: ABEL microsampler device — The ABEL microsampler device will be used to collect nasal fluid samples for biomarker analysis.

SUMMARY:
This research study is an observational, single site study quantifying expression of biomarkers of respiratory disease in nasal fluid using the ABEL microsampler device. The primary objective of this study is to compare biomarker expression between healthy controls and participants with respiratory disorders such as chronic obstructive pulmonary disorder (COPD), hayfever, chronic sinusitis, asthma and rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* All participants:
* 18 years of age or older
* The participant must be able to comprehend and sign an approved Informed Consent Form and other applicable study documents.
* Healthy volunteers:
* No significant sinonasal/pulmonary symptoms or prior diagnoses of sinonasal/pulmonary conditions as determined by pre-enrolment questionnaires.
* Case goup:
* Participants must be previously diagnosed with rhinitis, chronic sinusitis, asthma, or COPD by a medical professional.

Exclusion Criteria:

* Less than 18 years of age at the time of enrolment.
* Volunteers who are actively pregnant
* Prior history of adverse reaction or contraindicated to diagnostic testing including fingerprick blood sampling, pulmonary testing, nasal swab/sampling.
* Any other conditions limiting the volunteer's ability to complete study requirements in the judgement of the investigator/clinician
* Any nasal anatomical issue or finding which may limit the safe insertion of the ABEL collection device, as determined by investigator/clinician
* History of nasal surgery or trauma within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any individual aged 18+, either as a healthy control or a medically diagnosed sufferer of hayfever, asthma, rhinitis, chronic rhinosinusitis or chronic obstructive pulmonary disorder.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Nasal biomarker discovery | From participant enrollment to the end of the site visit (up to a maximum of 26 weeks)
  To establish a correlation between nasal molecular biomarkers and disease severity and quality of life in patients with respiratory conditions (rhinitis, chronic sinusitis, asthma, COPD) compared to healthy controls, aiming to develop an objective biomarker-based disease severity score.

SECONDARY OUTCOMES:
ABEL microsampler validation | For the duration of nasal fluid sample collection at the study site visit (2 hour site visit, with up to 20 minutes allocated for nasal fluid collection with breaks).
  To validate the tolerability and performance of the ABEL nasal microsampling device in collecting nasal fluids from patients with respiratory conditions and healthy controls. This evaluation will focus on assessing the user comfort, the ease of administration and the consistency and precision of sample collection.

CONTACTS AND LOCATIONS:
Locations (1):
- Diag-Nose Medical, Notting Hill, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsor website — https://diag-nose.io